CLINICAL TRIAL: NCT05237778
Title: The Nightmare Catcher: Modulating Dreams With Targeted Memory Reactivation
Brief Title: Combined Treatment of Nightmares With Targeted Memory Reactivation and Imagery Rehearsal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Lampros Perogamvros, Senior Clinical Fellow, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-02270
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Nightmares, REM-Sleep Type

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMR group (Experimental): Patients will receive a sound while they generate a positive outcome of imagery rehearsal therapy (IRT). They will also receive the sound during REM sleep.
  Interventions: Behavioral: Imagery Rehearsal Therapy and Targeted memory reactivation during REM sleep
- Control group (Active Comparator): Patients will not receive a sound while they generate a positive outcome of imagery rehearsal therapy (IRT). They will receive the same sound as the experimental group during REM sleep under the same conditions.
  Interventions: Behavioral: Imagery Rehearsal Therapy

INTERVENTIONS:
Behavioral: Imagery Rehearsal Therapy and Targeted memory reactivation during REM sleep — Emerging evidence shows that REM sleep plays a causal role in extinction learning, emotion regulation and consolidation of emotionally positive memories. By using targeted memory reactivation (TMR), a known method where we associate a sound with a waking experience (i.e., a positive outcome of imagery rehearsal therapy in this study) and strengthening it during REM sleep, we want to accelerate the remission of nightmares.
  Arms: TMR group
Behavioral: Imagery Rehearsal Therapy — These patients will receive the classic treatment of Imagery Rehearsal Therapy (IRT) for nightmares without any association with a sound.
  Arms: Control group

SUMMARY:
With this protocol, investigators examine whether targeted memory reactivation (TMR), a technique used to strengthen memories, can accelerate remission of nightmare disorder. This protocol uses TMR during REM sleep to strengthen positive memories generated by Imagery Rehearsal Therapy (IRT), a recommended treatment of nightmares. Patients with nightmare disorder are asked to perform an initial IRT session and, while they generate a positive outcome of their recurrent nightmare, half of the patients are exposed to a sound (TMR group), while no such pairing with a sound takes place for the other half (control group). During the next two weeks, all patients perform IRT every evening at home and are exposed to the sound during REM sleep with a wireless headband, which automatically detects sleep stages. Clinical evaluation of the severity of nightmares before and after (2-weeks follow-up and 3-months follow-up) this intervention takes place using the validated Nightmare Frequency Questionnaire (NFQ, primary outcome measure), which retrospectively identifies the frequency of nightmares. We hypothesize that patients treated with IRT and who are exposed, during REM sleep and over 14 nights, to a sound that had previously been associated with the new positive dream scenario of IRT (TMR group), will have more reduced frequency of nightmares compared to participants with stimulation of the same, but non-associated, sound during REM sleep (control group).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nightmare disorder according to the International Classification of Sleep Disorders (ICSD-3) diagnostic and coding manual
* Patients with at least moderate severity (>1 episode per week)

Exclusion Criteria:

* severe depression
* insomnia disorder
* psychosis or anxiety disorder
* other sleep disorder (e.g.,obstructive sleep apnea syndrome, restless legs syndrome)
* neurological disease
* use of medications that would be likely to produce nightmares (e.g. hypnotics, β-blockers, amphetamines, antimicrobial agents)
* use of anxiolytics, antipsychotic or antidepressant medication were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Nightmare Frequency Questionnaire (NFQ) | 2 weeks
  Validated self-report scale to assess the number of nightmares per week
Nightmare Frequency Questionnaire (NFQ) | 3 months
  Validated self-report scale to assess the number of nightmares per week

SECONDARY OUTCOMES:
Nightmare Distress Questionnaire (NDQ) | 2 weeks
  Validated self-report scale to assess the emotional disturbance attributed to the nightmares
Beck Depression Inventory (BDI-II) | 2 weeks
  Validated self-report scale to assess depressive symptoms
Pittsburgh Sleep Quality Index (PSQI) | 2 weeks
  Validated self-report scale to assess the quality of sleep
Proportion of the emotion 'joy' in dreams | 2 weeks
  Use of a dream diary
Proportion of the emotion 'fear' in dreams | 2 weeks
  Use of a dream diary
Nightmare Distress Questionnaire (NDQ) | 3 months
  Validated self-report scale to assess the emotional disturbance attributed to the nightmares
Beck Depression Inventory (BDI-II) | 3 months
  Validated self-report scale to assess depressive symptoms
Pittsburgh Sleep Quality Index (PSQI) | 3 months
  Validated self-report scale to assess the quality of sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sleep Medicine, University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No